CLINICAL TRIAL: NCT00340444
Title: Genetic Study of Inflammatory Bowel Disease
Brief Title: Genetic Studies of Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904045; 04-HG-N045
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-19

CONDITIONS: Inflammatory Bowel Disease
Keywords: Linkage; Covariates; Association; Fine Mapping; Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

SUMMARY:
This study will examine the existence of genetic regions that are believed to bring about a risk for inflammatory bowel disease (IBD), with its subtypes of Crohn's disease and ulcerative colitis. It will identify the locations of chromosomes responsible for hereditary IBD through linkage analysis, a technique in genetic research in which the occurrence of a disorder in a family is evaluated alongside a known genetic disorder. The project will also do fine mapping of genes and examine possible genes associated with IBD.

IBD is a chronic and often disabling disorder of the gastrointestinal tract, affecting about 500,000 Americans. Both Crohn's disease and ulcerative colitis share many characteristics, such as abdominal pain, bloody diarrhea, fever, fatigue, and malnutrition. But the main factors that distinguish these subtypes depend on the location and depth of inflammation. Tests and analyses can generally pinpoint some of the differences between the two, but sometimes there are major overlaps in characteristics, and the diagnosis is known as indeterminate IBD. The exact cause of IBD is not known, but genetic and environmental factors are known to contribute to risk for the disease. The single most important environmental risk factor has been smoking exposure at the time the diagnosis is made. Also, several genetic risk factors are ethnicity, family history, and polymorphisms-abilities to take on different forms-in the NOD2 gene.

Patients who have a diagnosis of IBD and their family members 5 years of age and older who have or do not have that diagnosis may be eligible for this study.

Participants will be asked to complete a questionnaire on their health, ethnic background, religion, habits, family medical history, and medications. Information will also be sought on the diagnosis, course, complications, and treatment of IBD, as well as risk factors. In addition, there will be collection of blood to be used for DNA preparation, storage of lymphocytes, and information on immunology.

DETAILED DESCRIPTION:
Using epidemiological, statistical, and molecular genetic techniques, this proposal is designed to investigate the existence of genetic regions that are believed to confer a risk for inflammatory bowel disease (IBD), which consists of two subtypes, Crohn's disease (CD) and ulcerative colitis (UC). The project will derive its study population, consisting of IBD physician confirmed affected probands with their family members, from the Johns Hopkins University, the University of Chicago, and the University of Pittsburgh. The project will consist of multiple parts. The first part is a reanalysis of existing genome wide linkage data from IBD families with 377 genotyped microsatellite marker data that incorporates covariate data into the analysis, with the goal of identifying new and refining previously identified regions of linkage. Eventually this may be extended to include new families typed for genome wide scan markers. The second part of the project consists of the fine mapping of the IBD3 locus (HLA region on chromosome 6p), which has been shown to have evidence of linkage in UC patients. Fifty-two microsatellite markers spanning the affected child trios in an effort to identify potential marker alleles that may be associated with UC, using the IBD3 locus will be genotyped in a study population consisting of 240 UC father-mother-affected child trios in an effort to identify potential marker alleles that may be associated with UC, using the transmission disequilibrium test, and to identify potential haplotypes that may confer an increased risk of developing UC, using a likelihood-based approach where a moving window of adjacent markers will be tested for excessive transmission. Additional candidate genes within IBD3 will be examined, and polymorphisms will also be tested for potential significant associations. Eventually this second part may be extended to fine mapping and association analysis of other candidate genes and/or candidate regions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants who have a diagnosis of IBD and their family members who have or do not have a diagnosis of IBD will be recruited for this study. Those further selected to be included in the linkage study must have at least two affected family members who are willing to donate blood samples and to fill out medical questionnaires.

EXCLUSION CRITERIA:

Children who were under the age of 5 years were excluded from the Johns Hopkins University recruitment protocol. There was no age restriction for the University of Chicago or the University of Pittsburgh. Those who were not able to provide consent were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000
Dates: Start 2003-11-06; Study Completion 2007-09-19

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Lee KS, Medline A, Shockey S. Indeterminate colitis in the spectrum of inflammatory bowel disease. Arch Pathol Lab Med. 1979 Apr;103(4):173-6. PMID 581845